CLINICAL TRIAL: NCT03106779
Title: A Phase 3, Multi-center, Open-label, Randomized Study of Oral ABL001 Versus Bosutinib in Patients With Chronic Myelogenous Leukemia in Chronic Phase (CML-CP), Previously Treated With 2 or More Tyrosine Kinase Inhibitors
Brief Title: Study of Efficacy of CML-CP Patients Treated With ABL001 Versus Bosutinib, Previously Treated With 2 or More TKIs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CABL001A2301; 2016-002461-66 (EudraCT Number)
Record Dates: First submitted 2017-03-09; First posted 2017-04-10 (Actual); Results first posted 2022-02-15 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Chronic Myelogenous Leukemia
Keywords: Phase 3; Chronic Myelogenous Leukemia; CML; bosutinib; ABL001; tyrosine kinase inhibitor; Chronic myelogenous leukemia (CML); chronic myeloid leukemia (CML); chronic myelocytic leukemia (CML); chronic granulocytic leukemia (CGL); cancer of the white blood cells; clonal bone marrow stem cell disorder; proliferation of mature granulocytes
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — asciminib; bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Asciminib (Experimental): Patients were randomized to asciminib 40mg BID
  Interventions: Drug: Asciminib
- Bosutinib (Active Comparator): Patients were randomized to bosutinib 500mg QD
  Interventions: Drug: Bosutinib

INTERVENTIONS:
Drug: Asciminib — 40 mg tablets was taken orally twice a day (BID)
  Other Names: ABL001
  Arms: Asciminib
Drug: Bosutinib — 500 mg tablets was taken orally once daily (QD)
  Arms: Bosutinib

SUMMARY:
The purpose of this pivotal study was to compare the efficacy of asciminib (ABL001) with that of bosutinib in the treatment of patients with CML-CP having previously been treated with a minimum of two prior ATP-binding site TKIs.

Patients intolerant to the most recent TKI therapy must have had BCR-ABL1 ratio > 0.1% IS at screening and patients failing their most recent TKI therapy must have met the definition of treatment failure as per the 2013 European LeukemiaNet (ELN) recommendations.

Patients with documented treatment failure as per 2013 ELN recommendations while on bosutinib treatment had the option to switch to asciminib treatment within 96 weeks after the last patient has been randomized on study.

DETAILED DESCRIPTION:
Patients were randomized in a 2:1 ratio to asciminib 40 mg BID or bosutinib 500 mg QD. Randomization was stratified by major cytogenetic response (MCyR) at screening. Patients with documented treatment failure (specifically meeting lack of efficacy criteria adapted from the 2013 ELN recommendations) while on bosutinib treatment were offered the option to switch to asciminib treatment within 96 weeks after the last patient was randomized to the study.

ELIGIBILITY:
Inclusion Criteria:

Male or female patients with a diagnosis of CML-CP ≥ 18 years of age

Patients must meet all of the following laboratory values at the screening visit:

* < 15% blasts in peripheral blood and bone marrow
* < 30% blasts plus promyelocytes in peripheral blood and bone marrow
* < 20% basophils in the peripheral blood
* ≥ 50 x 109/L (≥ 50,000/mm3) platelets
* Transient prior therapy related thrombocytopenia (< 50,000/mm3 for ≤ 30 days prior to screening) is acceptable
* No evidence of extramedullary leukemic involvement, with the exception of hepatosplenomegaly

BCR-ABL1 ratio > 0.1% IS according to central laboratory at the screening examination for patients intolerant to the most recent TKI therapy

Prior treatment with a minimum of 2 prior ATP-binding site TKIs (i.e. imatinib, nilotinib, dasatinib, radotinib or ponatinib)

Failure (adapted from the 2013 ELN Guidelines Bacarrani 2013) or intolerance to the most recent TKI therapy at the time of screening

* Failure is defined for CML-CP patients (CP at the time of initiation of last therapy) as follows. Patients must meet at least 1 of the following criteria.
* Three months after the initiation of therapy: No CHR or > 95% Ph+ metaphases
* Six months after the initiation of therapy: BCR-ABL1 ratio > 10% IS and/or > 65% Ph+ metaphases
* Twelve months after initiation of therapy: BCR-ABL1 ratio > 10% IS and/or > 35% Ph+ metaphases
* At any time after the initiation of therapy, loss of CHR, CCyR or PCyR
* At any time after the initiation of therapy, the development of new BCR-ABL1 mutations which potentially cause resistance to study treatment
* At any time after the initiation of therapy, confirmed loss of MMR in 2 consecutive tests, of which one must have a BCR-ABL1 ratio ≥ 1% IS
* At any time after the initiation of therapy, new clonal chromosome abnormalities in Ph+ cells: CCA/Ph+
* Intolerance is defined as:
* Non-hematologic intolerance: Patients with grade 3 or 4 toxicity while on therapy, or with persistent grade 2 toxicity, unresponsive to optimal management, including dose adjustments (unless dose reduction is not considered in the best interest of the patient if response is already suboptimal)
* Hematologic intolerance: Patients with grade 3 or 4 toxicity (absolute neutrophil count [ANC] or platelets) while on therapy that is recurrent after dose reduction to the lowest doses recommended by manufacturer

Exclusion Criteria:

Known presence of the T315I or V299L mutation at any time prior to study entry Known second chronic phase of CML after previous progression to AP/BC Previous treatment with a hematopoietic stem-cell transplantation Patient planning to undergo allogeneic hematopoietic stem cell transplantation

Cardiac or cardiac repolarization abnormality, including any of the following:

* History within 6 months prior to starting study treatment of myocardial infarction (MI), angina pectoris, coronary artery bypass graft (CABG)
* Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia), complete left bundle branch block, high-grade AV block (e.g., bifascicular block, Mobitz type II and third degree AV block)
* QTcF at screening ≥450 msec (male patients), ≥460 msec (female patients)
* Long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:
* Risk factors for Torsades de Pointes (TdP) including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia
* Concomitant medication(s) with a known risk of Torsades de Pointes per www.crediblemeds.org that cannot be discontinued or replaced 7 days prior to starting study drug by safe alternative medication.
* Inability to determine the QTcF interval
* Severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol (e.g. uncontrolled diabetes, active or uncontrolled infection, pulmonary hypertension)
* History of acute pancreatitis within 1 year of study entry or past medical history of chronic pancreatitis
* History of acute or chronic liver disease
* Treatment with medications that meet one of the following criteria and that cannot be discontinued at least one week prior to the start of treatment with study treatment
* Moderate or strong inducers of CYP3A
* Moderate or strong inhibitors of CYP3A
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 3 days after last dose of ABL001 and one month after last dose of bosutinib. Highly effective contraception methods include:
* Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
* Female sterilization (have had surgical bilateral oophorectomy (with or without hysterectomy) total hysterectomy or bilateral tubal ligation at least six weeks before taking study treatment). In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
* Male sterilization (at least 6 months prior to screening). The vasectomized male partner should be the sole partner for that subject.
* Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS) or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
* In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.
* Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or bilateral tubal ligation at least six weeks before taking study medication. In the case of oophorectomy alone, women are considered post-menopausal and not of child bearing potential only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2024-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (85):
- United States (10):
  - University of Chicago Hospital, Chicago, Illinois
  - Indiana Blood and Marrow Institute, Beech Grove, Indiana
  - Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Center, Boston, Massachusetts
  - University of Michigan Clinical Trials Office, Ann Arbor, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Cornell Medicine NY-Presb, New York, New York
  - Memorial Sloan Kettering Cancer Ctr, New York, New York
  - Uni Of TX MD Anderson Cancer Cntr, Houston, Texas
  - Utah Huntsman Cancer Center, Salt Lake City, Utah
- Argentina (3):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Capital Federal
  - Novartis Investigative Site, Córdoba
- Australia (3):
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Murdoch, Western Australia
- Brazil (3):
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Porto Alegre
- Bulgaria (2):
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Varna
- Novartis Investigative Site, Toronto, Ontario, Canada
- Czechia (2):
  - Novartis Investigative Site, Ostrava, Poruba
  - Novartis Investigative Site, Brno-Bohunice
- France (5):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Germany (7):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Kiel
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
- Israel (2):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Ẕerifin
- Italy (3):
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Napoli
- Japan (10):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Toyoake, Aichi-ken
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Ōsaka-sayama, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Chūō, Yamanashi
  - Novartis Investigative Site, Akita
  - Novartis Investigative Site, Aomori
  - Novartis Investigative Site, Kobe
- Lebanon (2):
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, El Achrafiyé
- Novartis Investigative Site, Monterrey, Nuevo León, Mexico
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Dordrecht
- Romania (2):
  - Novartis Investigative Site, Cluj-Napoca
  - Novartis Investigative Site, Timișoara
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Novartis Investigative Site, Riyadh, Saudi Arabia
- Serbia (2):
  - Novartis Investigative Site, Belgrade
  - Novartis Investigative Site, Novi Sad
- South Korea (4):
  - Novartis Investigative Site, Uijeongbu-si, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Jeollanam
- Spain (5):
  - Novartis Investigative Site, Bilbao, Basque Country
  - Novartis Investigative Site, Toledo, Castille-La Mancha
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Zurich, Switzerland
- Turkey (Türkiye) (5):
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Samsun
- United Kingdom (5):
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Mauro MJ, Minami Y, Hochhaus A, Lomaia E, Voloshin S, Turkina A, Kim DW, Apperley JF, Cortes JE, Abdo A, Fogliatto LM, Kim DDH, le Coutre P, Saussele S, Annunziata M, Hughes TP, Chaudhri N, Chee L, Garcia-Gutierrez V, Sasaki K, Boquimpani C, Kapoor S, Espurz N, Dhamal V, Rea D. Asciminib remained superior vs bosutinib in late-line CML-CP after nearly 4 years of follow-up in ASCEMBL. Blood Adv. 2025 Aug 26;9(16):4248-4259. doi: 10.1182/bloodadvances.2025016042. PMID 40334072
- [Derived] Cortes JE, Rea D, Mauro MJ, Tran D, Wang P, Jadhav K, Yocolly A, Sasaki K. Health care resource utilization in 3L + patients with chronic phase chronic myeloid leukemia receiving asciminib or bosutinib. J Med Econ. 2023 Jan-Dec;26(1):915-923. doi: 10.1080/13696998.2023.2234776. PMID 37431294
- [Derived] Yuda J, Doki N, Matsuoka H, Yokota T, Tomita A, Takahashi N, Matsumura I, Kubo K, Goto T, Kirito K, Maki A, Aoki M, Allepuz A, Minami Y. Asciminib vs bosutinib in CML patients pretreated with >/=2 tyrosine kinase inhibitors: Results from the Japanese subgroup analysis of ASCEMBL study. Cancer Med. 2023 Feb;12(3):2990-2998. doi: 10.1002/cam4.5212. Epub 2022 Sep 27. PMID 36168187
- [Derived] Li YF, Combes FP, Hoch M, Lorenzo S, Sy SKB, Ho YY. Population Pharmacokinetics of Asciminib in Tyrosine Kinase Inhibitor-Treated Patients with Philadelphia Chromosome-Positive Chronic Myeloid Leukemia in Chronic and Acute Phases. Clin Pharmacokinet. 2022 Oct;61(10):1393-1403. doi: 10.1007/s40262-022-01148-9. Epub 2022 Jun 28. PMID 35764773
- [Derived] Rea D, Mauro MJ, Boquimpani C, Minami Y, Lomaia E, Voloshin S, Turkina A, Kim DW, Apperley JF, Abdo A, Fogliatto LM, Kim DDH, le Coutre P, Saussele S, Annunziata M, Hughes TP, Chaudhri N, Sasaki K, Chee L, Garcia-Gutierrez V, Cortes JE, Aimone P, Allepuz A, Quenet S, Bedoucha V, Hochhaus A. A phase 3, open-label, randomized study of asciminib, a STAMP inhibitor, vs bosutinib in CML after 2 or more prior TKIs. Blood. 2021 Nov 25;138(21):2031-2041. doi: 10.1182/blood.2020009984. PMID 34407542

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 220 patients were planned to be enrolled, and 233 patients (157 randomized to treatment with asciminib and 76 to treatment with bosutinib) were enrolled and analyzed
Pre-assignment Details: Randomization was stratified by major cytogenetic response (MCyR) at screening.
Groups:
- Asciminib: Patients randomized to asciminib 40mg BID
- Bosutinib: Patients randomized to bosutinib 500mg QD
Period: Overall Study
Arm/Group | Asciminib | Bosutinib
Started | 157 | 76
Treated | 156 | 0
Not Treated (One patient randomized to asciminib was discontinued due to cytopenia as per Investigator's decision and never took medication.) | 1 | 0
Completed (Completed = Patients ongoing at the time of the primary analysis cut-off) | 97 | 22
Not Completed | 60 | 54
Not completed — Lack of Efficacy | 33 | 24
Not completed — Adverse Event | 8 | 16
Not completed — Physician Decision | 10 | 6
Not completed — Patient/guardian decision | 4 | 3
Not completed — Progressive disease | 1 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Death | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Not treated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): The FAS comprised of all randomized patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Asciminib | Bosutinib | Total
Number analyzed (Participants) | 157 | 76 | 233
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (13.49) | 51.0 (13.95) | 51.0 (13.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 45 | 120
  Male | 82 | 31 | 113
Race/Ethnicity, Customized [Number; unit: participants]
  White | 118 | 56 | 174
  Asian | 22 | 11 | 33
  Black or African American | 8 | 2 | 10
  American Indian or Alaska Native | 1 | 0 | 1
  Other | 5 | 7 | 12
  Unknown | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Molecular Response (MMR) Rate at 24 Weeks
Description: MMR was defined as a ≥ 3.0 log reduction in BCR-ABL1 transcripts compared to the standardized baseline equivalent to ≤ 0.1% BCR-ABL1/ABL% by IS as measured by RQ-PCR.
Time Frame: 24 weeks
Population: Full Analysis Set (FAS): The FAS comprised of all randomized patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Asciminib | Bosutinib
Number analyzed (Participants) | 157 | 76
Participants | 40 | 10
Statistical Analysis 1: Comparison: Asciminib vs Bosutinib; Test type: Superiority; p = 0.029, Cochran-Mantel-Haenszel; Stratified by the randomization stratification factor, i.e. cytogenetic response status (MCyR vs no MCyR) at screening; treatment difference in the MMR rate = 12.2, 95% CI 2-sided [2.19 to 22.30]

2. Secondary Outcome: Number of Participants With Major Molecular Response (MMR) Rate
Description: To compare additional parameters of the efficacy asciminib versus bosutinib
Time Frame: 96 weeks after the last patient received the first study dose
Reporting Status: Not Posted, anticipated posting 2025-12

3. Secondary Outcome: Complete Cytogenetic Response Rate
Description: To compare additional parameters of the efficacy of asciminib versus bosutinib. Cytogenic response will include Complete, Partial, Major, Minor, Minimal and no response.
Time Frame: 96 weeks after the last patient received the first study dose
Reporting Status: Not Posted, anticipated posting 2025-12

4. Secondary Outcome: Time to MMR
Description: To compare additional parameters of the efficacy of asciminib versus bosutinib
Time Frame: 96 weeks after the last patient received the first study dose
Reporting Status: Not Posted, anticipated posting 2025-12

5. Secondary Outcome: Duration of MMR
Description: To compare additional parameters of the efficacy of asciminib versus bosutinib
Time Frame: 96 weeks after the last patient received the first study dose
Reporting Status: Not Posted, anticipated posting 2025-12

6. Secondary Outcome: Time to CCyR
Description: To compare additional parameters of the efficacy of asciminib versus bosutinib
Time Frame: 96 weeks after the last patient received the first study dose
Reporting Status: Not Posted, anticipated posting 2025-12

7. Secondary Outcome: Duration of CCyR
Description: To compare additional parameters of the efficacy of asciminib versus bosutinib
Time Frame: 96 weeks after the last patient received the first study dose
Reporting Status: Not Posted, anticipated posting 2025-12

8. Secondary Outcome: Time to Treatment Failure
Description: To compare additional parameters of the efficacy of asciminib versus bosutinib
Time Frame: 96 weeks after the last patient received the first study dose
Reporting Status: Not Posted, anticipated posting 2025-12

9. Secondary Outcome: Progression Free Survival
Description: To compare additional parameters of the efficacy of asciminib versus bosutinib
Time Frame: 96 weeks after the last patient received the first study dose
Reporting Status: Not Posted, anticipated posting 2025-12

10. Secondary Outcome: Overall Survival
Description: To compare additional parameters of the efficacy of asciminib versus bosutinib
Time Frame: 96 weeks after the last patient received the first study dose
Reporting Status: Not Posted, anticipated posting 2025-12

11. Secondary Outcome: Trough Plasma Concentrations
Description: To characterize the PK of asciminib in the CML-CP population
Time Frame: 96 weeks after the last patient received the first study dose
Reporting Status: Not Posted, anticipated posting 2025-12

12. Secondary Outcome: PK Parameter: Cmax,
Description: To characterize the PK of asciminib in the CML-CP population
Time Frame: 96 weeks after the last patient received the first study dose
Reporting Status: Not Posted, anticipated posting 2025-12

13. Secondary Outcome: PK Parameter: Tmax
Description: To characterize the PK of asciminib in the CML-CP population
Time Frame: 96 weeks after the last patient received the first study dose
Reporting Status: Not Posted, anticipated posting 2025-12

14. Secondary Outcome: PK Parameter: AUC0-12h
Description: To characterize the PK of asciminib in the CML-CP population
Time Frame: 96 weeks after the last patient received the first study dose
Reporting Status: Not Posted, anticipated posting 2025-12

15. Secondary Outcome: PK Parameter: CL/F
Description: To characterize the PK of asciminib in the CML-CP population
Time Frame: 96 weeks after the last patient received the first study dose
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: For this interim results, Adverse Events were reported from informed consent (maximum 21 days before randomization) until end of treatment plus 30 days. The maximum duration of treatment exposure was 129.9 weeks for asciminib and 117 weeks for bosutinib.
Description: Adverse Event (AE): Any sign or symptom that occurs during treatment plus 30 days after study treatment discontinuation.
  Adverse events were analyzed in the Safety analysis set, which comprises all patients who received at least one dose of study treatment.
Arm/Group | Asciminib | Bosutinib
All-Cause Mortality (participants affected / at risk) | 4/156 | 1/76
Serious Adverse Events (participants affected / at risk) | 21/156 | 14/76
Other Adverse Events (participants affected / at risk) | 122/156 | 69/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Asciminib (N=156) | Bosutinib (N=76)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Toxic optic neuropathy (Eye disorders) | 1 | 0
Mesenteric artery embolism (Gastrointestinal disorders) | 1 | 0
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Hyperthermia (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
COVID-19 (Infections and infestations) | 1 | 0
Mycobacterium avium complex infection (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Device malfunction (Product Issues) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Angiopathy (Vascular disorders) | 1 | 0
Aortic occlusion (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Asciminib (N=156) | Bosutinib (N=76)
Anaemia (Blood and lymphatic system disorders) | 15 | 6
Neutropenia (Blood and lymphatic system disorders) | 28 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 35 | 10
Abdominal pain (Gastrointestinal disorders) | 7 | 11
Abdominal pain upper (Gastrointestinal disorders) | 7 | 5
Constipation (Gastrointestinal disorders) | 8 | 4
Diarrhoea (Gastrointestinal disorders) | 18 | 54
Dyspepsia (Gastrointestinal disorders) | 8 | 3
Nausea (Gastrointestinal disorders) | 18 | 35
Vomiting (Gastrointestinal disorders) | 11 | 19
Asthenia (General disorders) | 9 | 1
Fatigue (General disorders) | 16 | 7
Oedema peripheral (General disorders) | 9 | 2
Pyrexia (General disorders) | 4 | 6
Nasopharyngitis (Infections and infestations) | 15 | 2
Upper respiratory tract infection (Infections and infestations) | 10 | 4
Alanine aminotransferase increased (Investigations) | 6 | 21
Amylase increased (Investigations) | 9 | 4
Aspartate aminotransferase increased (Investigations) | 6 | 16
Lipase increased (Investigations) | 8 | 5
Neutrophil count decreased (Investigations) | 7 | 4
Platelet count decreased (Investigations) | 10 | 4
Decreased appetite (Metabolism and nutrition disorders) | 6 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 5
Dizziness (Nervous system disorders) | 10 | 2
Headache (Nervous system disorders) | 25 | 10
Insomnia (Psychiatric disorders) | 8 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 5
Rash (Skin and subcutaneous tissue disorders) | 11 | 17
Hypertension (Vascular disorders) | 18 | 3

LIMITATIONS AND CAVEATS:
In the asciminib arm, 2 patients died on-treatment and 2 patients died during survival follow-up. In the bosutinib arm, 1 patient died on-treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-14): https://cdn.clinicaltrials.gov/large-docs/79/NCT03106779/Prot_SAP_001.pdf